CLINICAL TRIAL: NCT02589119
Title: A Phase I Study of Autologous Mesenchymal Stromal Cell Coated Fistula Plug in Patients With High, Transsphincteric Cryptoglandular Perianal Fistulas
Brief Title: Stem Cell Fistula Plug in Cryptoglandular Perianal Fistulas (MSC-AFP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Eric J. Dozois, M.D., MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-003200
Record Dates: First submitted 2015-10-21; First posted 2015-10-28 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Perianal Fistula; Cryptoglandular Perianal Fistula
Keywords: cryptoglandular; perianal fistula; cryptoglandular perianal fistulas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSC-AFP (Other): Single Treatment Group
  Interventions: Drug: MSC-AFP

INTERVENTIONS:
Drug: MSC-AFP — Eligible patients will be treated with a fistula plug that has been coated with autologous mesenchymal stromal cell.
  Other Names: mesenchymal stromal cell coated fistula plug

SUMMARY:
The investigators propose to study the safety of autologous mesenchymal stromal cell transfer using a biomatrix (the Gore Fistula Plug) in a Phase I study using a single dose of 20 million cells. 15 adult patients, ages 18 years and older with cryptoglandular fistulas will be enrolled. Subjects will undergo standard adjuvant therapy including drainage of infection and placement of a draining seton. Six weeks post placement of the draining seton, the seton will be replaced with the MSC loaded Gore Fistula Plug; fistula plug as per current clinical practice. The subjects will be subsequently followed for fistula response and closure for 24 months. This is an autologous product derived from the patient and used only for the same patient.

DETAILED DESCRIPTION:
The investigators propose to study the safety of autologous mesenchymal stromal cell transfer using a biomatrix (the Gore® Bio-A® Fistula Plug) in a Phase I study using a single dose of 20 million cells. 15 adult patients (age > 18 years) with cryptoglandular fistulas will be enrolled. Subjects will undergo standard adjuvant therapy including drainage of infection and placement of a draining seton. Six weeks post placement of the draining seton, the seton will be replaced with the MSC loaded Gore® fistula plug as per current clinical practice. The subjects will be subsequently followed for fistula response and closure for 24 months. Study visits are Day 1, Week 2, Week 4, Week 8, Week 12, Week 24, Week 52, and Week 104. This is an autologous product derived from the patient and used only for the same patient.

ELIGIBILITY:
Inclusion Criteria

1. Males and females 18-65 years of age.
2. Residents of the United States.
3. Single-tract, transsphincteric anal fistula of cryptoglandular origin. Primary fistulas (no previous surgical treatment) and those who have failed previous surgical repairs
4. Have no contraindications to MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia
5. Ability to comply with protocol
6. Competent and able to provide written informed consent

Exclusion Criteria

1. Inability to give informed consent.
2. Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
3. Specific exclusions; Evidence of hepatitis B, C, or HIV
4. History of cancer including melanoma (with the exception of localized skin cancers)
5. Investigational drug within thirty (30) days of baseline
6. A resident outside the United States
7. Pregnant or breast feeding.
8. History of clinically significant auto-immunity (e.g. Crohn's disease) or any previous example of fat-directed autoimmunity
9. Previous allergic reaction to a perianal fistula plug.
10. If liposuction is not technically feasible
11. Allergic to local anesthetics
12. Pregnant patients or trying to become pregnant.
13. Non-enterocutaneous tracts (i.e. recto-vaginal, entero-vesicular)
14. Multi-tract, suprasphincteric and extrasphincteric fistula tract extensions
15. Active local infection associated with the fistula

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (safety and toxicity). | 2-24 months
  Participants will have a health assessment and blood work measured at each study visit to monitor for adverse events, such as worsening of the cryptoglandular fistulizing disease, abnormal laboratory values, or significant abnormalities in physical examination. The Outcome Measure will be the number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment

SECONDARY OUTCOMES:
Number of participants with response to the treatment regarding potential cessation of drainage from their fistula. | 2-24 months
  Participants will have a clinical assessment of fistula drainage. Participants will be assessed during an office examination if their fistula is draining or not. The Outcome Measure will be the presence or absence of fistula drainage.

OTHER OUTCOMES:
Number of participants with response to the treatment regarding their score based on the Cleveland Clinic Florida (Wexner) fecal incontinence questionnaire. | 6-12 months
  Participants will have an assessment with the Cleveland Clinic Florida (Wexner) fecal incontinence questionnaire. Participants have the questionnaire administered within one week before plug implantation and at the 6 month and 12 months follow up visits. The Outcome Measure will be the how the participants' score change over time.
Number of participants with radiographic healing response to the treatment. | 2-24 months
  Participants will have an assessment of healing radiographically by magnetic resonance imaging (MRI). Participants' fistula tracts will be assessed during a MRI if their fistula is healing. The Outcome Measure will be the closure or persistence of fistula tract.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Dozois, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials